CLINICAL TRIAL: NCT04752813
Title: A Study of BPM31510 With Vitamin K1 in Subjects With Newly Diagnosed Glioblastoma (GB)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BPGbio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPM31510IV-11
Record Dates: First submitted 2021-02-01; First posted 2021-02-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Vitamin K 1; Temozolomide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BPM31510, Vitamin K1, RT and TMZ (Experimental): Subjects will receive a BPM31510 96hr infusion once weekly for 8 wk. Prophylactic Vitamin K1 at a recommended dose of 10 mg will be given subcutaneously to all subjects prior to the beginning of each week of therapy.
  After 2 wk of treatment with BPM31510, subjects will start concurrent standard RT and TMZ 75 mg/m2 once daily (qd) × 42 days. Subjects will receive the standard TMZ treatment for up to 12 cycles post BPM31510 treatment.
  Interventions: Drug: BPM31510; Other: Vitamin K1; Drug: Temozolomide (TMZ); Radiation: Radiation

INTERVENTIONS:
Drug: BPM31510 — Subjects will receive a weekly, 96-h infusion of BPM31510 for a duration of 8 weeks.
Other: Vitamin K1 — Subjects will receive prophylactic Vitamin K1 at a recommended dose of 10 mg subcutaneously prior to the beginning of each week of BPM31510 therapy.
Drug: Temozolomide (TMZ) — After 2 wk of treatment with BPM31510 (ie, on Day 15), subjects will start concurrent TMZ 75 mg/m2 once daily (qd) × 42 days. Subjects will receive the standard TMZ treatment for up to 12 cycles post BPM31510 treatment.
Radiation: Radiation — After 2 wk of treatment with BPM31510 (ie, on Day 15), subjects will start concurrent standard RT for 42 days.

SUMMARY:
This is a single-arm, non-randomized, open-label Phase 2 therapeutic study that will assess the effects of adding BPM31510 onto a conventional treatment framework of RT and concurrent TMZ chemotherapy for subjects with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
The study will start with a dose-confirmation phase to establish safety of BPM31510 in combination with RT and TMZ. This phase will follow a standard 3+3 dose design with the starting dose of BPM31510 at 110 mg/kg/week (wk), with 1 potential dose de-escalation to 66 mg/kg/wk in the event a DLT is experienced at the 110 mg/kg dose. Toxicity at this dose level will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5 (CTCAE v5). Subjects will be monitored for DLTs associated with combination therapy for 30 days (d) (± 5 d) after the end of RT (DLT assessment period). Subjects will continue to be monitored for late radiation-related DLTs during follow up, every 8 wk (± 2 wk) during the first 12 months (mo), and then every 12 wk (± 2 wk) for a total of 5 years (y). Safety oversight will be provided by the independent Data and Safety Monitoring Committee (DSMC). The DSMC will review and confirm all DLT data, make recommendations for dose modifications, if necessary, and continue to monitor safety throughout the study. The efficacy phase of the study will begin after the recommended Phase 2 dose (RP2D) has been confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with newly diagnosed pathologically verified GB.
2. No prior RT, chemotherapy, immunotherapy, or targeted agents administered specifically for the lesion being treated.
3. Age ≥18 y.
4. Life expectancy ≥3 months.
5. Karnofsky performance score ≥60.
6. Adequate organ and marrow function as per protocol.
7. Ability for subject to understand and the willingness to sign a written ICF.
8. Subjects of childbearing potential must agree to use hormonal or barrier birth control with spermicidal gel to avoid pregnancy during the study.
9. Be at least 15 d out and not more than 50 d from surgery.

Exclusion Criteria:

1. History of clinically significant tumor-related cerebral hemorrhage.
2. Patients with multicentric disease defined by tumors which have multiple discrete areas of contrast-enhancing tumor without connecting T2/FLAIR signal abnormality.
3. Patients with diffuse leptomeningeal disease.
4. Patients who are not eligible for definitive surgical resection.
5. Patients on decadron daily dosing more than 2 mg.
6. Any serious cardiac history as per protocol.
7. Uncontrolled or severe coagulopathies or a history of clinically significant bleeding within the past 6 months.
8. Known predisposition for bleeding such as von Willebrand's disease or other such condition(s).
9. Uncontrolled concurrent illness.
10. Prior malignancy except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 3 y prior to first dose of study drug.
11. Receiving any of the following medications:

    1. Therapeutic doses of any anticoagulant, including low-molecular weight heparin. Concomitant use of warfarin, even at prophylactic doses, is prohibited.
    2. Digoxin, digitoxin, lanatoside C, or any type of digitalis alkaloids.
    3. Antiangiogenic drugs (ie, Avastin) either in the past 2 wk or if anticipated within the next 2 wk of informed consent.
    4. Theophylline
12. Known allergy to CoQ10.
13. Known allergy or adverse reaction to Vitamin K1.
14. Pregnant or lactating.
15. Known to be positive for the human immunodeficiency virus (HIV). Note: HIV testing is not required for eligibility, but if performed previously and was positive, the subject is ineligible.
16. Patients with a contraindication to radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2030-08-26 (Estimated)

PRIMARY OUTCOMES:
Efficacy will be assessed by subject progression free survival | 6 months and 12 months
  Progression free survival will be determined by measuring the proportion of subjects who have met RANO criteria for complete response, partial response , or stable disease at 6 mo and 12 mo following initiation of BPM31510.

SECONDARY OUTCOMES:
Efficacy will be assessed by subject Overall survival | 5 years
  Overall survival as determined by measuring from start date of BPM31510 to the date of death or date of last follow-up (for subjects who have not died).
Safety and tolerability of BPM31510 and Vitamin K1 will be assessed by incidence of dose limiting toxicities (DLTs) and adverse events (AEs). | 30 days post treatment
  A DLT is defined as an event possibly related to BPM31510 and clearly not due to an underlying disease or extraneous causes. An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Cancer Center, Palo Alto, California
  - Sansum Clinic, Santa Barbara, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Valley Health, Ridgewood, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Texas Oncology, Austin, Texas
  - UT Health San Antonio Mays Cancer Center, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Inova, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia